CLINICAL TRIAL: NCT00872339
Title: Assessment of Pain in People With Thalassemia
Acronym: Pain
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 639; U01HL065238 (NIH)
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-01

CONDITIONS: Thalassemia
Keywords: Transfusion-Dependent Thalassemia; Non-Transfusion-Dependent Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- transfusion-dependant: People with transfusion-dependant thalassemia who received at least 8 transfusions in the past year.
- non-transfusion-dependant: People with non-transfusion-dependant thalassemia who received no transfusions in the past year.
- intermittently transfused: Intermittently transfused patients- individuals who received at least one but fewer than eight transfusions in the last year

SUMMARY:
Thalassemia is an inherited blood disorder that can result in mild to severe anemia. People with thalassemia often experience pain, but the exact sources and prevalence of pain remain unknown. This study will examine the prevalence and severity of pain in people with thalassemia who are treated with regular blood transfusions and people with thalassemia who are not treated with regular blood transfusions.

DETAILED DESCRIPTION:
Thalassemia is an inherited blood disorder in which the body makes an abnormal form of hemoglobin-the protein in red blood cells that carries oxygen. People with thalassemia often experience fatigue, shortness of breath, and pain. Recent medical advances in treating people with thalassemia who receive regular blood transfusions-a standard procedure that refreshes the healthy red blood supply-have resulted in increased life spans for these people. However, with the extended life spans have come additional issues, including pain. There have been no previous research studies that have examined pain levels in people with thalassemia, and as a result, the sources and prevalence of pain remain unknown. The purpose of this study is to assess the prevalence and severity of pain, common pain sites, and the impact of pain on functioning and well-being in people with thalassemia who receive regular blood transfusions and people with thalassemia who do not receive regular blood transfusions.

This study will enroll people with transfusion-dependant thalassemia and people with non-transfusion-dependant thalassemia. At a baseline study visit, participants will complete a demographic questionnaire and a pain assessment questionnaire. At Months 3, 6, and 9, study researchers will telephone participants to go over the same pain assessment questionnaire again.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia, as documented by clinical diagnosis, including the following:

  1. B-thalassemia (intermedia or major)
  2. Hgb H disease
  3. Hgb H with non-deletional mutations (e.g., Hgb H Constant Spring)
  4. E-B-thalassemia
  5. Homozygous alpha thalassemia
  6. Other thalassemic conditions not explicitly excluded
  7. Thalassemia intermedia due to heterozygous B mutation with an alpha excess
* Participants can be of any race, ethnicity, and either gender.

Exclusion Criteria:

* Thalassemia trait (i.e., single recessive B gene mutation, 2 gene alpha mutation) and thalassemia Hgb S, C, or D compound heterozygotes
* Unwillingness or inability to complete the Brief Pain Inventory (BPI) on a quarterly basis
* Has had a successful bone marrow transplant

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thalassemia patients who receive regular blood transfusions and those who do not receive regular blood transfusions.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Boudreeaux, MD, Principal Investigator — Children's Healthcare of Atlanta; Ellis Neufeld, MD, Principal Investigator — Boston Children's Hospital; Alexis Thompson, MD, Principal Investigator — Children's Memorial Hospital of Chicago; Brigitta Mueller, MD, Principal Investigator — Baylor College of Medicine at Houston; Dru Foote, RN, NP, Study Chair — Children's Hospital and Research Institute of Oakland; Patricia Giardina, MD, Principal Investigator — Weill Medical College of Cornell; Janet Kwiatkowski, MD, Principal Investigator — Children's Hospital of Philadelphia; Nancy Olivieri, MD, Principal Investigator — Toronto General Hospital
Locations (8):
- United States (7):
  - Children's Hospital and Research Institute at Oakland, Oakland, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Boston, Boston, Massachusetts
  - Weill Medical College, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Haines D, Martin M, Carson S, Oliveros O, Green S, Coates T, Eile J, Schilling L, Dinu B, Mendoza T, Gerstenberger E, Trachtenberg F, Vichinsky E; Thalassemia Clinical Research Network. Pain in thalassaemia: the effects of age on pain frequency and severity. Br J Haematol. 2013 Mar;160(5):680-7. doi: 10.1111/bjh.12177. Epub 2012 Dec 30. PMID 23278768

RESULTS

PARTICIPANT FLOW:
Groups:
- Transfusion-dependant: People with transfusion-dependant thalassemia.
- Intermittently Transfused: Intermittently transfused patients- individuals who received fewer than eight transfusions in the last year
- Non-transfusion-dependant: People with non-transfusion-dependant thalassemia.
Period: Overall Study
Arm/Group | Transfusion-dependant | Intermittently Transfused | Non-transfusion-dependant
Started | 201 | 14 | 37
Completed | 201 | 14 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transfusion-dependant | Intermittently Transfused | Non-transfusion-dependant | Total
Number analyzed (Participants) | 201 | 14 | 37 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (10.4) | 35.8 (14.4) | 29.5 (16.2) | 28.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 6 | 14 | 137
  Male | 84 | 8 | 23 | 115

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Pain
Time Frame: Measured at Month 9
Measure: Number; unit: participants
Arm/Group | Transfusion-dependant | Intermittently Transfused | Non-transfusion-dependant
Number analyzed (Participants) | 201 | 14 | 37
participants | 75 | 7 | 11
Statistical Analysis 1: Comparison: Transfusion-dependant vs Intermittently Transfused vs Non-transfusion-dependant; Test type: Superiority or Other; p = 0.45, Chi-squared

2. Secondary Outcome: Common Sites of Pain
Time Frame: Measured at Month 9
Measure: Number; unit: participants
Groups:
- All Subjects Combined: Subjects with pain in the last 7 days were combined into one group.
Arm/Group | All Subjects Combined
Number analyzed (Participants) | 93
participants
  Lower back | 76
  Either leg | 52
  Head | 45
  Midback | 44
  Either hip | 36
  Upper back | 36
  Either arm | 29
  Abdomen | 26
  Chest | 25

3. Secondary Outcome: Pain Occurrence by Age
Time Frame: Measured at Month 9
Measure: Number; unit: participants
Groups:
- All Subjects Combined: Subjects were combined into one group.
Arm/Group | All Subjects Combined
Number analyzed (Participants) | 252
participants
  12-17 yo (n=50) | 4
  18-24 (n=56) | 19
  25-34 (n=61) | 22
  35-44 (n=61) | 34
  45-71 (n=24) | 14
Statistical Analysis 1: Comparison: All Subjects Combined; Test type: Superiority or Other; p < .001, Chi-squared

4. Secondary Outcome: Impact of Pain on Functioning and Well-being
Time Frame: Measured at Month 9
Measure: Number; unit: participants
Arm/Group | All Subjects Combined
Number analyzed (Participants) | 93
participants
  Mood | 83
  Normal work | 76
  General activities | 74
  Sleep | 74
  Walking | 73
  Enjoyment of life | 69
  Interpersonal relations | 57

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Groups:
- Adverse Events Were Not Collected: Adverse events were not collected for this study.
Arm/Group | Adverse Events Were Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No